CLINICAL TRIAL: NCT02823587
Title: Effects of Pulmonary Rehabilitation on Secretion Transport, Inflammation and Respiratory System Strength and Quality of Life in Patients With Bronchiectasis
Brief Title: Pulmonary Rehabilitation in Non-Cystic Fibrosis Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USP 2016-1
Record Dates: First submitted 2016-05-19; First posted 2016-07-06 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2016-12

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Mucociliary clearance; Exercise; Inflammation
MeSH Terms: conditions — Bronchiectasis; Motor Activity; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bronchiectasis Pulmonary Rehabilitation (Experimental): The volunteers will receive supervised physical training twice a week and will be instructed to adopt a routine of home exercises, for 12 weeks.
  Interventions: Other: Pulmonary Rehabilitation
- Healthy Pulmonary Rehabilitation (Experimental): In this arm, the volunteers healthy will receive supervised physical training twice a week and will be instructed to adopt a routine of home exercises, for 12 weeks.
  Interventions: Other: Pulmonary Rehabilitation
- Bronchiectasis Group Control (Sham Comparator): The volunteers with bronchiectasis will be informed only about the benefits of physical activities
  Interventions: Other: Control
- Healthy Group Control (Sham Comparator): Volunteers healthy will be informed only about the benefits of physical activities
  Interventions: Other: Control

INTERVENTIONS:
Other: Pulmonary Rehabilitation — The exercise program will consist of an individual exercise prescription on the treadmill or bike, the initial intensity of 85% VO2max and active exercises or active-resistance for upper and lower limbs according to the capacity of each volunteer.
  Arms: Bronchiectasis Pulmonary Rehabilitation; Healthy Pulmonary Rehabilitation
Other: Control — No supervised exercise session, only will be informed at the beginning of the study to perform thirty minutes of physical activity of moderate intensity several days a week is associated with health benefits
  Arms: Bronchiectasis Group Control; Healthy Group Control

SUMMARY:
The purpose of this study is to assess the effect of pulmonary rehabilitation on the transport of secretions, inflammation and respiratory resistance, and its repercussions on the quality of life in patients with bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is characterized by pathological and irreversible dilation of bronchi caused by the inefficient removal of secretions and microorganisms and the perpetuation of inflammatory processes induced by chronic or recurrent infections, causing more damage to the airways that result in infections, and greater lesion airways and lung parenchyma. Pulmonary rehabilitation in people with bronchiectasis aims to improve exercise capacity, through effects on aerobic capacity and peripheral muscles, and to improve disease control and quality of life. The aim this study is to evaluate the effects of pulmonary rehabilitation on the transport of secretions, inflammation and respiratory resistance, and its repercussions on the quality of life in patients with bronchiectasis. In this study 60 volunteers, of both sexes, aged between 18-60 years, adequate the inclusion criteria, which will be assessed by lung function tests, the saccharin transport time, the inflammatory markers in the airways, the respiratory system resistance and quality of life scales. Volunteers will be randomly divided in pulmonary rehabilitation (PRG) and control groups (CG) that will be subdivided in bronchiectasis and healthy subgroups. In the PRG group they will receive supervised physical training twice a week and will be instructed to adopt a routine of home exercises, while CG will be informed about the benefits of physical activities. All volunteers will be evaluated after 8 weeks of the baseline and at the end of the research. Data evolution will be collected from medical records and notes of the medical team and physical therapy that will follow the routine of these participants

ELIGIBILITY:
Inclusion Criteria:

* clinically stable patients
* both sexes
* aged between 18-60 years
* not due to cystic fibrosis bronchiectasis diagnosis
* non smokers
* no pulmonary disease

Exclusion Criteria:

* asthma or other restrictive conditions
* smokers assets
* decompensated cardiovascular and metabolic diseases, neuromuscular or musculoskeletal that impede the realization of the Protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mucociliary transport in vivo | Through study completion, an average of 2 years.
  This measurement it will be evaluated by the saccharine transport time, according to methodology (Stanley, 1984)

SECONDARY OUTCOMES:
Mucociliary transport in vitro | Through study completion, an average of 2 years.
  This measurement it will be evaluated by the transport properties in vitro, according to methodology (Trindade, 1997)
Quality of Life in Bronchiectasis | Through study completion, an average of 2 years.
  For this evaluation the investigators will use the Quality of life in bronchiectasis (QOLB) (Chalmers, 2014)
Cough Impact Assessment | Through study completion, an average of 2 years.
  For this evaluation the investigators will use the Leicester Cough Questionnaire (LCQ), (Murray, 2009).
Health-Related Quality of Life | Through study completion, an average of 2 years.
  For this evaluation the investigators will use the Short Form Health Survey (SF-36) (Ware, 1992)
Impulse Oscillometry System (IOS) | Through study completion, an average of 2 years.
  To perform this measure, it is been used Jaeger® IOS(Jaeger, Wurzburg, Germany) with daily volume and resistance calibration. The parameters are calculated at frequencies between 5 and 35 hertz, and will be analyzed the following parameters in this test: resistance (R), reactance (X), reactance area (AX) and resonant frequency (Fres).
Pulmonary Function Test | Through study completion, an average of 2 years.
  This test is realized by using KoKo Spirometer™ according American Thoracic Society (ATS)/European Respiratory Society (ATS)recommendations. The analyzed parameters in this test are: forced vital capacity (FVC), Forced Expiratory Volume in the First Second (FEV1), FEV1/FVC and forced expiratory flow (FEF25-75%).
Six Minute Walking Test | Through study completion, an average of 2 years.
  Patients walk through a 30 meter corridor faster than they can for 6 minutes, according to ATS considerations.
Maximal Static Respiratory Pressures | Through study completion, an average of 2 years.
  It has beem used a digital manometer (MVD300, Global Med, São Paulo, Brazil) with graduation ranging from 0 to ± 300 centimeters of water (cmH2O) and adjusted to a rigid mouthpiece, following the proposed model by Black and Hyatt in 1969.
Viscosity | Through study completion, an average of 2 years.
  To perform this measure, it is been used a capillary viscometer dual-chamber is used for measuring viscosity of bronchial mucus (Barnett et al, 1970)
Elasticity | Through study completion, an average of 2 years.
  To perform this measure, it is been used a capillary viscometer dual-chamber is used for measuring elasticity of bronchial mucus (Kim, 1988)
Exhaled breath condensate | Through study completion, an average of 2 years
  It will be collected as previously described (Koczulla et al., 2009).
Exhaled Nitric Oxide Fraction (FeNO) | Through study completion, an average of 2 years
  It will be performed according to protocol defined by the American Thoracic Society (ATS, 2011), using the device NioxMino™.
Cytokine Analysis TNF-α | Through study completion, an average of 2 years
  The tumor necrosis factor-alpha concentrations (TNF-α) in the nasal lavage fluid(NFL) (samples will be determined using immunohistochemistry high sensitivity assays(ELISA), which will be performed according to the instructions the kit supplier.
Cytokine Analysis IL-6 | Through study completion, an average of 2 years
  The interleukins(IL) - IL-6 in the NFL samples will be determined using immunohistochemistry high sensitivity assays(ELISA), which will be performed according to the instructions the kit supplier.
Cytokine Analysis IL-10 | Through study completion, an average of 2 years
  The interleukins - IL-10 in the NFL samples will be determined using immunohistochemistry high sensitivity assays(ELISA), which will be performed according to the instructions the kit supplier.

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PhD, Principal Investigator — Ribeirão Preto Medicine School - University of São Paulo
Locations (1):
- Ribeirão Preto Medical School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Stanley P, MacWilliam L, Greenstone M, Mackay I, Cole P. Efficacy of a saccharin test for screening to detect abnormal mucociliary clearance. Br J Dis Chest. 1984 Jan;78(1):62-5. PMID 6691910
- [Background] Mandal P, Sidhu MK, Kope L, Pollock W, Stevenson LM, Pentland JL, Turnbull K, Mac Quarrie S, Hill AT. A pilot study of pulmonary rehabilitation and chest physiotherapy versus chest physiotherapy alone in bronchiectasis. Respir Med. 2012 Dec;106(12):1647-54. doi: 10.1016/j.rmed.2012.08.004. Epub 2012 Sep 1. PMID 22947443
- [Background] Trindade SH, de Mello JF Jr, Mion Ode G, Lorenzi-Filho G, Macchione M, Guimaraes ET, Saldiva PH. Methods for studying mucociliary transport. Braz J Otorhinolaryngol. 2007 Sep-Oct;73(5):704-12. doi: 10.1016/s1808-8694(15)30133-6. PMID 18094814
- [Background] Koczulla R, Dragonieri S, Schot R, Bals R, Gauw SA, Vogelmeier C, Rabe KF, Sterk PJ, Hiemstra PS. Comparison of exhaled breath condensate pH using two commercially available devices in healthy controls, asthma and COPD patients. Respir Res. 2009 Aug 24;10(1):78. doi: 10.1186/1465-9921-10-78. PMID 19703285